CLINICAL TRIAL: NCT04301934
Title: Fractional CO2 Vaginal LASER Therapy for Recurrent Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johnny Yi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-002297
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Estrogens, Conjugated (USP); Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vaginal Estrogen Therapy Group (Active Comparator): Women randomized to vaginal estrogen therapy will be offered vaginal cream conjugated estrogen (Premarin) 0.5 gm per vaginal twice weekly or estradiol (Estrace): 1gm per vaginal twice weekly
  Interventions: Drug: Conjugated estrogen; Drug: Estradiol
- Laser Therapy Group (Experimental): Women randomized to the laser therapy group will undergo 3 treatments, 6 weeks apart.
  Interventions: Device: Mona Lisa Touch

INTERVENTIONS:
Device: Mona Lisa Touch — Fractional CO2 LASER
  Arms: Laser Therapy Group
Drug: Conjugated estrogen — Current standard treatment for recurrent UTIs in postmenopausal women
  Other Names: Premarin
  Arms: Vaginal Estrogen Therapy Group
Drug: Estradiol — Current standard treatment for recurrent UTIs in postmenopausal women
  Other Names: Estrace
  Arms: Vaginal Estrogen Therapy Group

SUMMARY:
Randomized controlled trial to determine clinical and microbiome difference between fractional CO2 Laser and vaginal estrogen in treating patients with recurrent urinary tract infection (UTI).

DETAILED DESCRIPTION:
Recurrent urinary tract infection (rUTI) is common in postmenopausal women and can lead to significant bothersome symptoms. This clinical scenario is a difficult and common clinical problem seen by the urologist and urogynecologist with limited options for treatment. Overuse of antibiotics has led to significant resistant microorganisms and can have adverse side effects such as C. Dificile colitis. Current treatments include topical vaginal estrogen and prophylactic antibiotics. Other supplements such as cranberry pills, methenamine and D-mannose have varying levels of evidence and efficacy.

Fractional CO2 LASER vaginal therapy has recently been studied for the treatment of GSM. LASER therapy is currently commercially available and has FDA clearance for use in gynecology. Current evidence shows that with treatment, histologic changes of the vaginal epithelium have shown regeneration to a premenopausal state, along with subjective improvement in GSM symptoms and sexual function. Recent literature has shown improvements in thickening of vaginal epithelium, decreased vaginal pH and improvement in the vaginal microbiome. Based on this, the investigators propose fractional CO2 laser may have a positive impact on women with rUTI.

1. The investigators therefore hypothesize that fractional CO2 LASER vaginal therapy is non-inferior to topical vaginal estrogen therapy for the treatment of rUTI.

   a. Primary Outcome: Improvement in recurrence of culture positive UTI
2. The investigators also hypothesize that LASER therapy will improve the urinary and vaginal microbiome, decreasing the uropathogenic presence and increasing Lactobacillus.

   1. Measurement 1: The number of UTI with UPEC isolated from patients
   2. Measurement 2: The pH of the vagina as a proxy for presence of Lactobacillus sp.
   3. Measurement 3: Categorize vaginal and urinary microbial communities
3. The investigators hypothesize that LASER therapy will improve symptoms of GSM and be associated with regenerative change in vaginal histology.

   1. Measurement 1: MESA and DIVA surveys of symptoms
   2. Measurement 2: Observations of vaginal biopsy between.

Menopausal women will be recruited if subjects have recurrent UTI defined as 3 culture positive UTIs in 1 year or 2 culture positive UTIs in 6 months. Subjects will be randomized to standard of care with topical vaginal estrogen or 3 treatments of fractional CO2 LASER of the vagina. Samples will be collected to show microbiome and histologic changes with treatment.

Samples include:

Vaginal culture Urine culture vaginal biopsy (optional).

Validated questionnaires and clinical recurrence of UTI will also be gathered over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patient >18 years old
* Postmenopausal status, documented by prior bilateral salpingo-oophorectomy, or absence of menses >12 months
* Recurrent urinary tract infections as defined by 3 culture positive urine cultures in the last 12 months, or 2 positive urine cultures in the last 6 months.(Positive urine cultures defined by >100K colony forming units of 1 or 2 bacterial species on clean catch sample, or >1000 colony forming units of 1 or 2 bacterial species on sample via straight catheterization).
* Patients on vaginal estrogen must undergo a 1 month washout period prior to initiation of the trial.

Exclusion Criteria:

* Hematuria without appropriate workup
* Pelvic organ prolapse at or beyond the hymen
* Clinically relevant urinary retention
* Pelvic reconstructive surgery within 6 months
* Prior synthetic mesh procedure for pelvic organ prolapse or urinary incontinence
* Clinically relevant nephrolithiasis
* History of breast cancer
* Contraindication to topical estrogen therapy
* Anticoagulation therapy
* Prior pelvic or vaginal radiation therapy
* Prior gynecologic malignancy
* Undiagnosed genital bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Yi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaginal Estrogen Therapy Group: Women randomized to vaginal estrogen therapy were offered vaginal cream conjugated estrogen (Premarin) 0.5 gm per vaginal twice weekly or estradiol (Estrace): 1gm per vaginal twice weekly
  Conjugated estrogen: Current standard treatment for recurrent UTIs in postmenopausal women
  Estradiol: Current standard treatment for recurrent Urinary Tract Infections (UTI) in postmenopausal women
- Laser Therapy Group: Women randomized to the laser therapy group underwent 3 treatments, 6 weeks apart.
  Mona Lisa Touch: Fractional CO2 LASER
Period: Overall Study
Arm/Group | Vaginal Estrogen Therapy Group | Laser Therapy Group
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vaginal Estrogen Therapy Group: Women randomized to vaginal estrogen therapy were offered vaginal cream conjugated estrogen (Premarin) 0.5 gm per vaginal twice weekly or estradiol (Estrace): 1gm per vaginal twice weekly
  Conjugated estrogen: Current standard treatment for recurrent UTIs in postmenopausal women
  Estradiol: Current standard treatment for recurrent UTIs in postmenopausal women
- Total: Total of all reporting groups
Arm/Group | Vaginal Estrogen Therapy Group | Laser Therapy Group | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (6.41) | 69.1 (9.47) | 68.0 (7.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Urinary Tract Infections (UTI)
Description: Prevalence of urinary tract infections (UTI) described as percentage of subjects with none vs one or more UTI.
Time Frame: 4 months
Measure: Number; unit: percentage of subjects
Arm/Group | Vaginal Estrogen Therapy Group | Laser Therapy Group
Number analyzed (Participants) | 7 | 5
percentage of subjects
  No UTI | 28.6 | 60
  1 + UTI | 71.4 | 40
Statistical Analysis 1: Comparison: Vaginal Estrogen Therapy Group vs Laser Therapy Group; Test type: Non-Inferiority — The prevalence of UTI for the LASER group and vaginal estrogen group was calculated. Non-inferiority test using Farrington-Manning method was applied to test the risk difference against the pre-specified non-inferiority margin (20%); p = 0.034, Farrington-Manning

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 6 months
Arm/Group | Vaginal Estrogen Therapy Group | Laser Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/5
Other Adverse Events (participants affected / at risk) | 3/7 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Estrogen Therapy Group (N=7) | Laser Therapy Group (N=5)
Urospepsis with positive urine and blood cultures (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Estrogen Therapy Group (N=7) | Laser Therapy Group (N=5)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal irritation (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Abnormal bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (5)
Increase vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal burning (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vaginal itching (Reproductive system and breast disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04301934/Prot_SAP_000.pdf